CLINICAL TRIAL: NCT02078180
Title: Pharmacokinetic Study of Bupropion Hydrochloride Products With Different Release Patterns
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Duxin Sun, Professor of Pharmaceutical Sciences, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HHSF223201310164C; HUM00081894 (Other: UM IRBMED)
Record Dates: First submitted 2014-02-28; First posted 2014-03-05 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Bupropion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- generic bupropion IR75 (Active Comparator): One oral dose of generic bupropion IR75
  Interventions: Drug: generic bupropion
- generic bupropion IR100 (Active Comparator): One oral dose of generic bupropion IR100
  Interventions: Drug: generic bupropion
- generic bupropion SR100 (Active Comparator): One oral dose of generic bupropion SR100
  Interventions: Drug: generic bupropion
- generic bupropion SR150 (Active Comparator): One oral dose of generic bupropion SR150
  Interventions: Drug: generic bupropion
- generic bupropion XL150 (Active Comparator): One oral dose of generic bupropion XL150
  Interventions: Drug: generic bupropion
- generic bupropion XL300 (Active Comparator): One oral dose of generic bupropion XL300
  Interventions: Drug: generic bupropion

INTERVENTIONS:
Drug: generic bupropion — We are comparing different formulations of bupropion that release this drug at different rates. The abbreviation IR75 means immediate release and the number is the dose in mg. The other abbreviations represent SR for sustained-release and XL for extended release, which release the drug slower than the IR formulation.
  Other Names: Wellbutrin

SUMMARY:
The objectives of this project are to determine if the bioavailability and release pattern of bupropion HCl products differ and if the genotype of the metabolic enzymes affects the saturation of intestinal enzymes with different dose strengths within one product line. Findings from this project will help the FDA Center for Drug Evaluation and Research's (CDER) Office of Generic Drugs improve policy development and review practice in the future for similar products, e.g. extended release oral drug products being metabolized in the gut wall and having multiple strengths.

Aim 1: To compare the pharmacokinetics of bupropion and its metabolites in plasma in healthy individuals when they ingest different strengths of bupropion (75-300 mg) with variable release profiles (IR vs XL vs SR) in GI tract.

Working hypothesis: Variation in release rate and mechanism of bupropion formulations in gastrointestinal (GI) tract will impact metabolism and saturation of bupropion in GI tract, which will generate different concentration of bupropion and its metabolites in plasma.

Aim 2: To investigate pharmacogenomics of CYP 2B6 that influences metabolism, saturation, and pharmacokinetics of bupropion

Working hypothesis: The gain of function of CYP2B6 variants (allele *4 and *22) in patients will increase the metabolism of bupropion in the GI tract and liver, reduce both local concentration and plasma concentration of bupropion, and thus cause non-bioequivalence when bupropion is released earlier in GI tract

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers 25 to 55 years old.
* Volunteers have a Body Mass Index (BMI), calculated from the ratio of height and weight, within a range of 18.5 to 35.
* Willing to be medication and supplement free 2 weeks prior to beginning study, and throughout the study. All forms of birth control are okay.

Exclusion Criteria:

* Individuals unwilling or unable to comply with the study protocol (e.g. unable to remain medication or supplement free during the study).
* Individuals unwilling or unable to take bupropion or have an allergy to bupropion
* Any medical or surgical conditions which might significantly alter bupropion absorption (e.g., history of malabsorption, liver disease, gastric bypass surgery )
* Individuals with a history of psychiatric or neurological illness, including seizure disorders
* Nicotine dependence
* Alcohol dependence
* Pregnant or nursing women

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2014-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duxin Sun, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IR75, IR200, SR100, SR150, XL150, XL300: Participants were randomized to receive one pill each of IR 75, IR 100, SR 100, SR 150, XL 150 and XL 300,in randomized order at six time points. Given the large number of possible sequence combinations, participants are reported as a single Participant Flow Arm with Milestones used to indicate how many participants received each intervention
Period: Overall Study
Arm/Group | IR75, IR200, SR100, SR150, XL150, XL300
Started | 34
IR75 | 30
IR100 | 31
SR100 | 31
SR150 | 32
XL 150 | 31
XL 300 | 32
Completed | 29
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- IR 75, IR 100, SR 100, SR 150, XL 150 and XL 300: Participants were randomized to receive one pill each of IR 75, IR 100, SR 100, SR 150, XL 150 and XL 300,in randomized order at six time points. Given the large number of possible sequence combinations, participants are reported as a single Participant Flow Arm with Milestones used to indicate how many participants received each intervention
Arm/Group | IR 75, IR 100, SR 100, SR 150, XL 150 and XL 300
Number analyzed (Participants) | 34
Age, Customized [Count of Participants; unit: Participants]
  <25 years | 0
  25-65 years | 34
  >65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 24
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Comparision of the Buproprion Area Under the Concentration Time Curve (AUC) From Time 0 to 96 Hours by Type of Formulation and Dosage
Description: Each formulation of buproprion has a different rate of release. Some release the drug immediately while others release the drug slowly. We will compare the exposure of buproprion by formulation and dose by looking at the area under the concentration time curve. The area under the concentration time curve is a mathematical way of looking at drug exposure in the body. The reported values are AUC (0-96 hours).
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: h*nanogram/milliliter
Arm/Group | Generic Bupropion IR75 | Generic Bupropion IR100 | Generic Bupropion SR100 | Generic Bupropion SR150 | Generic Bupropion XL150 | Generic Bupropion XL300
Number analyzed (Participants) | 30 | 31 | 30 | 32 | 30 | 30
h*nanogram/milliliter | 469 (177) | 667 (418) | 706 (304) | 1002 (516) | 740 (449) | 1356 (637)

2. Secondary Outcome: Comparision of the Buproprion Maximum Concentration (Cmax) by Type of Formulation and Dosage
Description: Each formulation of buproprion has a different rate of release. Some release the drug immediately while others release the drug slowly. We will compare the exposure of buproprion by formulation and dose by looking at the maximum concentration. The maximum concentration depends on the rate of drug release and so looking at this value can help us compare differences between formulation.
Time Frame: 4 days
Measure: Mean (Standard Error); unit: nanogram/milliliter
Arm/Group | Generic Bupropion IR75 | Generic Bupropion IR100 | Generic Bupropion SR100 | Generic Bupropion SR150 | Generic Bupropion XL150 | Generic Bupropion XL300
Number analyzed (Participants) | 30 | 31 | 30 | 32 | 30 | 30
nanogram/milliliter | 93 (36) | 136 (70) | 61 (29) | 78 (40) | 61 (34) | 111 (44)

ADVERSE EVENTS:
Time Frame: Varied per person from 3 months to 10 months based on their randomization sequence and the time that it took to complete all phases of the study with washout between each formulation.
Arm/Group | IR 75, IR 100, SR 100, SR 150, XL 150 and XL 300
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 10/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IR 75, IR 100, SR 100, SR 150, XL 150 and XL 300 (N=34)
Headache (Nervous system disorders) | 5 (5)
Peripheral vision loss (Eye disorders) | 1 (1) — Briefly experienced loss of peripheral vision in right eye for approximately 30 minutes 6 days after dose. Full vision came back and participant did not experience anything out of the ordinary before or since resolution of vision loss.
Nausea (Gastrointestinal disorders) | 2 (2)
Dizzyness (Nervous system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Rash on both arms following completion of phase six of the study. Rash was located near site of blood draws on arms.

LIMITATIONS AND CAVEATS:
The small study sample size may have masked the contribution of pharmacogenetics to bupropion metabolism.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes